CLINICAL TRIAL: NCT00803023
Title: Safety and Tolerability Study Comparing Sodium Oxybate Given as an Oral Solution to a Single-blinded Combination of Oral Tablets Plus Oral Solution in Subjects With Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sr. Director of Clinical Development - Psychiatry, Jazz Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 08-004
Record Dates: First submitted 2008-12-03; First posted 2008-12-05 (Estimated); Results first posted 2011-08-16 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Sodium Oxybate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Sodium Oxybate Oral Solution (4.5 grams)
  Interventions: Drug: Sodium Oxybate
- 2 (Experimental): Sodium Oxybate taken as a combination of an Oral Solution and Placebo Tablets (4.5 grams)
  Interventions: Drug: Sodium Oxybate & 6 Tablets
- 3 (Experimental): Sodium Oxybate Oral Solution (6 grams)
  Interventions: Drug: Sodium Oxybate Oral Solution (6 grams)
- 4 (Experimental): Sodium Oxybate taken as a combination of an Oral Solution and Placebo Tablets (6 grams)
  Interventions: Drug: Sodium Oxybate & 8 Tablets

INTERVENTIONS:
Drug: Sodium Oxybate — 4.5 grams per night taken in two equally divided doses
  Arms: 1
Drug: Sodium Oxybate & 6 Tablets — 4.5 grams taken as a combination of liquid and 6 Placebo tablets in two equally divided doses per night
  Arms: 2
Drug: Sodium Oxybate & 8 Tablets — 6 grams taken as a combination of liquid and 8 Placebo tablets in two equally divided doses per night
  Arms: 4
Drug: Sodium Oxybate Oral Solution (6 grams) — 6 grams per night taken in two equally divided doses
  Arms: 3

SUMMARY:
To compare the safety and tolerability of sodium oxybate given as a combination of an oral solution and oral tablets for 4 weeks in subjects with fibromyalgia (FM).

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to understand the written informed consent
* Subject is 18 years of age or older.
* Subject meets the ACR criteria for fibromyalgia
* Subject is willing to discontinue prohibited by the protocol
* Subject agrees to use only non-sedating over-the-counter (OTC)medication
* Subject is willing to abstain from the ingestion of alcohol for the duration of the trial.

Exclusion Criteria:

* Subject has protocol prohibited medical & psychiatric conditions that would exclude subject
* Subject has a current or past history of a substance use disorder including alcohol abuse
* Subject has a clinically significant history of seizure disorder either past or present
* Female subject who is pregnant, nursing or lactating.
* Subject is diagnosed with sleep apnea
* Subject is unable to discontinue protocol prohibited medications
* Subject is experiencing fatigue and/or drowsiness/sedation in association with intake of allowed medications.
* Subject has taken any investigational drug within 5 half-lives of the investigational drug prior to signing the informed consent form.
* Subject has an allergic reaction to GHB or sodium oxybate or any of its constituents (e.g. malic acid).
* Subject is on a sodium-restricted diet.
* Subject has abnormal liver function test or other abnormal lab values
* Subject has an occupation that requires variable shift work or routine night shifts or cannot routinely spend at least 6 hours per night in bed.
* Subject has any other problems that, in the investigator's opinion, would preclude the subject's participation and completion of this trial or compromise reliable representation of subjective symptoms.
* Subject has been randomized into a previous Xyrem (sodium oxybate) clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace Wang, MD, Study Director — Jazz Pharmaceuticals
Locations (32):
- United States (32):
  - Dba 21st Century Neurology, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Orange County Clinical Trials, Anaheim, California
  - Med Investigations, Inc., Fair Oaks, California
  - Northridge Neurological Center, Northridge, California
  - Arroyo Medical Group, Inc., Pismo Beach, California
  - Northern California Research, Sacramento, California
  - Superior Research, LLC, Sacramento, California
  - Apex Research Institute, Santa Ana, California
  - Clinical Physiology Associates Clinical Study, Fort Meyers, Florida
  - Compass Research, Orlando, Florida
  - Memorial Medical Group - Clinical Research, South Bend, Indiana
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Commonwealth Biomedical Resaerch, LLC, Madisonville, Kentucky
  - Louisiana Sleep Foundation, Baton Rouge, Louisiana
  - Professional clinical Research - Interlochen, Interlochen, Michigan
  - Quality Clinical Research, Inc, Omaha, Nebraska
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Hill Top Physicians Inc. / Hihgtop Medical Research Center, Cincinnati, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Central Pennsylvania Clinic, Mechanicsburg, Pennsylvania
  - Southern Orthopeadic Sports, Columbia, South Carolina
  - The Carolina Center for Rheumatology & ArthiritisCare PA, Rock Hill, South Carolina
  - Clinsearch, Chattanooga, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - DFW Wellness, Fort Worth, Texas
  - Houston Sleep Clinic, Houston, Texas
  - Sun Research Institute, San Antonio, Texas
  - Clinical Health Research, LLC, Sugar Land, Texas
  - Pacific Rheumatology Associates, Renton, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- 4.5g SXB: Sodium Oxybate Oral Solution (4.5 grams/night)
- 4.5g SXB + 6 Tablets: Sodium Oxybate Oral Solution (4.5 grams/night)and 6 Placebo Tablets per night
- 6g SXB: Sodium Oxybate Oral Solution (6 grams/night)
- 6g SXB + 8 Tablets: Sodium Oxybate Oral Solution (6 grams/night) and 8 Placebo Tablets per night
Period: Overall Study
Arm/Group | 4.5g SXB | 4.5g SXB + 6 Tablets | 6g SXB | 6g SXB + 8 Tablets
Started | 32 | 33 | 31 | 33
Completed | 27 | 25 | 20 | 25
Not Completed | 5 | 8 | 11 | 8
Not completed — Adverse Event | 5 | 4 | 8 | 6
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 2 | 1
Not completed — Lack of Efficacy | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4.5g SXB | 4.5g SXB + 6 Tablets | 6g SXB | 6g SXB + 8 Tablets | Total
Number analyzed (Participants) | 32 | 33 | 31 | 33 | 129
Age Continuous [Mean (Standard Deviation); unit: years] | 48.3 (12.31) | 49.6 (11.69) | 49.3 (12.76) | 50.7 (12.24) | 49.5 (12.13)
Age, Customized [Number; unit: Participants]
  18 - 39 | 9 | 7 | 7 | 5 | 28
  40 - 49 | 6 | 6 | 8 | 8 | 28
  50 - 64 | 15 | 18 | 12 | 17 | 62
  >=65 | 2 | 2 | 4 | 3 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 27 | 32 | 119
  Male | 1 | 4 | 4 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 3 | 7 | 20
  Not Hispanic or Latino | 27 | 28 | 28 | 26 | 109
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 2 | 0 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 1 | 5
  White | 29 | 31 | 28 | 30 | 118
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 32 | 33 | 31 | 33 | 129

OUTCOME MEASURES:

1. Primary Outcome: Summary of Most Frequent Adverse Events (Per Arm) Experienced by Study Subjects
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | 4.5g SXB | 4.5g SXB + 6 Tablets | 6g SXB | 6g SXB + 8 Tablets
Number analyzed (Participants) | 32 | 33 | 31 | 33
participants
  Any Adverse Event | 20 | 21 | 21 | 23
  Gastrointestinal Disorders | 7 | 6 | 5 | 11
  Diarrhea | 0 | 0 | 1 | 2
  Nausea | 4 | 3 | 2 | 7
  Vomiting | 0 | 1 | 1 | 2
  General Disorders & Administration Site Conditions | 2 | 4 | 5 | 6
  Fatigue | 1 | 0 | 0 | 3
  Edema Peripheral | 1 | 2 | 1 | 1
  Infections & Infestation | 3 | 5 | 2 | 3
  Sinusitis | 0 | 1 | 1 | 2
  Urinary Tract Infection | 0 | 2 | 0 | 0
  Injury, Posioning, & Procedural Complications | 4 | 0 | 0 | 0
  Investigations | 0 | 3 | 3 | 1
  Metabolism & Nutrition Disorders | 0 | 0 | 3 | 1
  Musculoskeletal & Connective tissue Disorders | 2 | 3 | 3 | 3
  Back Pain | 1 | 0 | 2 | 2
  Nervous System Disorders | 8 | 5 | 9 | 10
  Dizziness | 3 | 1 | 4 | 2
  Headache | 2 | 3 | 2 | 3
  Somnolence | 0 | 0 | 1 | 2
  Tremor | 0 | 0 | 0 | 2
  Psychiatric Disorders | 4 | 5 | 5 | 11
  Anxiety | 1 | 1 | 0 | 2
  Insomnia | 2 | 3 | 0 | 3
  Major Depression | 1 | 0 | 2 | 0
  Renal & Urinary Disorders | 0 | 2 | 0 | 0
  Respiratory, Thoracic, & Mediastinal Disorders | 2 | 2 | 2 | 5
  Pharyngolaryngeal Pain | 0 | 1 | 0 | 2
  Sinus Congestion | 0 | 0 | 0 | 2
  Skin & Subcutaneous Tissue Disorders | 1 | 1 | 3 | 3

2. Secondary Outcome: Tolerability Assessed by Adverse Events
Time Frame: 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | 4.5g SXB | 4.5g SXB + 6 Tablets | 6g SXB | 6g SXB + 8 Tablets
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/33 | 1/31 | 0/33
Other Adverse Events (participants affected / at risk) | 12/32 | 13/33 | 11/31 | 17/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4.5g SXB (N=32) | 4.5g SXB + 6 Tablets (N=33) | 6g SXB (N=31) | 6g SXB + 8 Tablets (N=33)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal Behavior (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Major Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 4.5g SXB (N=32) | 4.5g SXB + 6 Tablets (N=33) | 6g SXB (N=31) | 6g SXB + 8 Tablets (N=33)
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 4 | 3 | 2 | 7
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Fatigue (General disorders) | 1 | 0 | 0 | 3
Edema Peripheral (General disorders) | 1 | 2 | 1 | 1
Sinusitus (Infections and infestations) | 0 | 1 | 1 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 2 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2
Dizziness (Nervous system disorders) | 3 | 1 | 4 | 2
Headache (Nervous system disorders) | 2 | 3 | 2 | 3
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 2
Tremor (Nervous system disorders) | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 3 | 0 | 3
Major Depression (Psychiatric disorders) | 1 | 0 | 2 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No